CLINICAL TRIAL: NCT00954109
Title: Physical Inactivity and Insulin Resistance in Skeletal Muscle
Brief Title: Acute Cardiovascular and Metabolic Effects of Exercise Training in Individuals With Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDA-2-051-07S; NCT00572676 (obsolete NCT alias)
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Insulin Resistance
Keywords: Insulin Resistance; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): exercise - supervised exercise (treadmill walking or cycle ergometer use)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — daily exercise: supervised treadmill walking or cycle ergometry use

SUMMARY:
The overall aim of the project is to determine whether or not exercise influences cardiovascular or nervous responses to meal ingestion in individuals with insulin resistance or type 2 diabetes.

DETAILED DESCRIPTION:
Participants will undergo a screening procedure, including telephone screening and physical examination, as well as determination of body composition and fitness. Participants will be asked to complete 5-10 days of supervised exercise training and will undergo testing to assess cardiovascular and metabolic responses to an oral glucose tolerance test, including muscle sympathetic nerve activity, blood flow, and circulating glucose and insulin concentrations at baseline and following training. In addition, day-to-day variations in blood glucose will also be monitored. The overall aim of the project is to determine whether or not acute exercise training influences postprandial metabolic, vascular or autonomic nervous system responses in individuals with insulin resistance or T2D.

ELIGIBILITY:
Inclusion Criteria:

* Insulin resistant: diagnosed with pre-diabetes or fasting blood glucose >/= 100 mg/dL
* T2D: diagnosed by primary care physician
* BMI: less than 43 kg/m2
* Age: 30-65

Exclusion Criteria:

* Smoking
* Insulin use (other than once daily)
* Underlying conditions that limit ability to exercise safely
* Recent weight gain or loss (>5% of body weight in 3 months)
* Physically active (>30 min aerobic exercise, 2 d/wk)
* Recent (<3 mo) changes in medication use or dose
* Uncontrolled T2D (HbA1c>10%)
* Advanced retinopathy or neuropathy
* Pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Thyfault, PhD, Principal Investigator — Harry S. Truman Memorial VA Medical Center
Locations (1):
- Harry S. Truman Memorial VA Medical Center, Columbia, Missouri, United States

REFERENCES:
- [Result] Mikus CR, Fairfax ST, Libla JL, Boyle LJ, Vianna LC, Oberlin DJ, Uptergrove GM, Deo SH, Kim A, Kanaley JA, Fadel PJ, Thyfault JP. Seven days of aerobic exercise training improves conduit artery blood flow following glucose ingestion in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Sep;111(3):657-64. doi: 10.1152/japplphysiol.00489.2011. Epub 2011 Jul 7. PMID 21737826
- [Derived] Mikus CR, Oberlin DJ, Libla J, Boyle LJ, Thyfault JP. Glycaemic control is improved by 7 days of aerobic exercise training in patients with type 2 diabetes. Diabetologia. 2012 May;55(5):1417-23. doi: 10.1007/s00125-012-2490-8. Epub 2012 Feb 4. PMID 22311420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: exercise - supervised exercise (treadmill walking or cycle ergometer use)
  Exercise: daily exercise: supervised treadmill walking or cycle ergometry use
Arm/Group | Arm 1
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity After 5-7 Days of Exercise
Description: Insulin sensitivity measured during an oral glucose tolerance test measured by the Matsuda Index. Matsuda insulin sensitivity index= 10000/square root of [(fasting glucose × fasting insulin) × (mean glucose × mean insulin during oral glucose tolerance test).
Time Frame: baseline and 24h after 5-7 days of exercise
Measure: Mean (Standard Error); unit: index score
Arm/Group | Arm 1
Number analyzed (Participants) | 11
index score
  Baseline | 3 (.2)
  Post 5-7 days of exercise | 2.5 (0.3)
Statistical Analysis 1: Comparison: Arm 1; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Primary Outcome: Blood Flow in Response to Oral Glucose Tolerance Tests
Description: Blood flow response in the femoral artery measured by Doppler ultrasound during and oral glucose tolerance test. Data are represented as % change in blood flow during the oral glucose tolerance at 60 minutes vs. 0 minutes (prior to drinking the glucose)
Time Frame: pre and 24 hours post 5-7 days of exercise
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Arm 1
Number analyzed (Participants) | 11
percentage change
  Baseline | 0 (2)
  Post 5-7 days of exercise | 40 (20)
Statistical Analysis 1: Comparison: Arm 1; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No